CLINICAL TRIAL: NCT04399954
Title: A Study to Evaluate the Acceptability of Ketoflo, a Food for Special Medical Purposes (FSMP) for Use in the Dietary Management of Epilepsy or Neurometabolic Conditions Requiring a Ketogenic Diet (KD)
Brief Title: Evaluation of Ketoflo
Acronym: Ketoflo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCT-KFLO-2018-02-19; 232386 (Other: IRAS); 19/NW/0018 (Other: HRA)
Record Dates: First submitted 2020-05-18; First posted 2020-05-22 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Epilepsy Intractable; Glucose Transporter Type 1 Deficiency Syndrome; Ketogenic Dieting
MeSH Terms: conditions — Drug Resistant Epilepsy; Glut1 Deficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Single group - all patients to receive Ketoflo.
Masking Description: No masking, product will be given open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketoflo (Experimental): Ketoflo to be incorporated into each participant's usual ketogenic diet for 28 days. Amount taken and frequency of intake to be determined by the dietitian.
  Interventions: Dietary Supplement: Ketoflo

INTERVENTIONS:
Dietary Supplement: Ketoflo — Ketoflo is a ready to use liquid feed for the dietary management of epilepsy and other conditions that may require a ketogenic diet. It has a 4:1 ratio of fat to carbohydrate and protein and can be administered enterally via a tube feeding or oral consumption.

SUMMARY:
For 28 days, 30 participants aged 3 to 18 years of age (inclusive) with a condition requiring a ketogenic diet will incorporate Ketoflo into their usual dietary regime. Ketoflo is a nutritionally complete Food For Special Medical Purposes and is suitable for administration by both tube feeding and use as a sip feed. Data on gastrointestinal tolerance, participants adherence to recommended intakes and their thoughts on the product's palatability will be self-reported in Daily Study Diaries.

DETAILED DESCRIPTION:
This is a 28-day prospective study to evaluate the acceptability of Ketoflo, in terms of GI tolerance, adherence to recommended intakes and palatability. The product's nutritional suitability for use in a ketogenic diet will also be evaluated by recording ketone levels and seizure frequency measured as part of usual clinical care.

Ketoflo is nutritionally complete liquid feed for use in the dietary management of epilepsy or other neurometabolic conditions requiring a ketogenic diet. It is designed to be nutritionally complete from 3-18 years and can be used as a supplementary feed thereafter.

Ketoflo has been designed in liaison with Key Opinion Leaders and will offer an additional choice of prescribe-able feeds for use in the ketogenic diet.

The study will involve 30 participants, aged between three and eighteen years of age (inclusive), who are already established on a ketogenic diet for at least three months before the study begins.

Participants will self-report data in Daily Study Diaries over the course of the study. Data will also be collected by the Investigators in Baseline CRFs and End of Study CRFs for all participants. Any data collected for the study will be anonymised before being relayed to the sponsor.

The data generated by the trial will be used to support a submission by Vitaflo (International) Ltd. to the Advisory Committee on Borderline Substances (ACBS) for Ketoflo to become reimbursable on prescription in the UK. The data will also be used in a submission to the General Medical Services in the Republic of Ireland.

ELIGIBILITY:
Inclusion Criteria:

i) Diagnosis of a condition requiring a ketogenic diet (KD) e.g. intractable epilepsy, Glut-1 deficiency syndrome (Glut-1 DS) etc.

ii) Aged 3 - 18 years of age (inclusive).

iii) Established on a ketogenic diet for at least 3 months under the supervision of a clinician and/or dietitian trained in the use of the KD.

iv) Requirement for a liquid ketogenic feed.

v) In the opinion of the investigator, the participant (and parent/guardian, if relevant) is/are able to comply with the study protocol requirements and complete the diary and questionnaire.

vi) Willingly given, written, informed consent from participant (or parent/guardian, if relevant)

vii) Willingly given, written assent (if appropriate).

Exclusion Criteria:

i) Inability to comply with the study protocol, in the opinion of the investigator.

ii) Under 3 years of age or over 18 years of age.

iii) Medical conditions in which the KD is contraindicated.

iv) Previous clinical evaluation indicating unsuitability for the KD.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in gastrointestinal tolerance from week 1 to week 4 | Days 1 - 7 and days 21 - 28.
  Participants will self-report any gastrointestinal symptoms experienced over the course of the study in Daily Study Diaries.
Adherence | Days 1 - 28.
  Participants will record the amount of Ketoflo taken each day compared to the amount recommended by their dietitian.
Palatability and ease of use | Day 28.
  Participants will answer questions relating to Ketoflo's palatability and ease of use following the end of the study.
Nutritional suitability: ketone levels | Days 1 - 28
  Ketoflo's nutritional suitability will be assessed by evaluating ketone levels (mmol/l) recorded by participants as part of routine care. These data will be recorded in the Daily Study Diaries.
Nutritional suitability: seizure frequency | Days 1 - 28
  Ketoflo's nutritional suitability will be assessed by evaluating seizure frequency (number per day) recorded by participants as part of routine care. These data will be recorded in the Daily Study Diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Lightfoot, Study Director — Leeds Teaching Hospitals NHS Trust
Locations (5):
- United Kingdom (5):
  - Royal Aberdeen Children's Hospital, Aberdeen
  - Barberry, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Leeds Children's Hospital, Leeds
  - Great Ormond Street Hospital for Children, London

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD.